CLINICAL TRIAL: NCT00217230
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial To Assess Safety And Efficacy Of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T) In Adults Aged 60 Years And Older CAIV-T, Liquid Formulation
Brief Title: Trial To Assess Safety And Efficacy Of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T) In Adults Aged 60 Years And Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D153-P507
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

INTERVENTIONS:
Biological: CAIV-T

SUMMARY:
The purpose of this study is to determine the efficacy, safety and tolerability of the liquid formulation of CAIV-T against culture confirmed influenza illness in adults aged 60 years and older. In addition this study aims to demonstrate superiority of CAIV-T when compared with placebo and the effect on economic resources.

DETAILED DESCRIPTION:
To evaluate the efficacy over 1 year against culture-confirmed influenza-illness caused by community-acquired subtypes antigenically similar to those contained in the vaccine, in adults aged ≥ 60 years at enrollment, of 1 dose of an intranasally-administered (IN) liquid formulation of influenza virus vaccine, trivalent, types A and B, live, cold-adapted (CAIV-T; Wyeth, Marietta, PA, USA) compared with saline placebo.

ELIGIBILITY:
Inclusion Criteria:

* who are and aged at least 60 years or older at the time of enrollment;
* who are determined by medical history, physical examination and clinical judgement to be eligible for this study. Subjects with stable pre-existing disease, defined as disease not requiring change in therapy or hospitalization within 12 weeks before receipt of study vaccination will be eligible.
* who have provided written informed consent after the nature of the study has been explained;
* who, will be available for duration of the trial (from enrollment to approximately November 30, 2001); who can be reached by study staff for the post-vaccination and weekly surveillance contacts [telephone, clinic or home visit].

Exclusion Criteria:

* who are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* who are a resident of a nursing home or long-term care facility or other institution receiving skilled or semi-skilled nursing care (refer to study manual). An ambulatory subject who is a resident of a retirement home or village is eligible for the trial.
* With evidence of dementia or other severe cognitive impairment based on Mini Mental State Examination (MMSE) scores (refer to study manual).
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; or cytotoxic agents;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* have an immunosuppressed or an immunocompromised individual living in the same household;
* with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine or placebo;
* who were administered any live virus vaccine within one month prior to enrollment or expected to receive another live virus vaccine within one month of vaccination in this study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* who, received a dose of influenza treatment (commercial or investigational) one month prior to enrollment. The prophylactic use of influenza antivirals is not permitted.
* who receive any influenza vaccine in the 6 months to enrollment, or a non-study influenza vaccine since enrollment;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results; Note: A pregnant household member is not considered a contraindication to enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2001-04; Study Completion 2001-11

PRIMARY OUTCOMES:
The primary study endpoint was the comparison of efficacy of CAIV-T versus placebo against culture-confirmed influenza-illness caused by community-acquired influenza subtypes that were antigenically similar to those contained in the vaccine.

SECONDARY OUTCOMES:
A secondary comparison of interest was the incidence of culture-confirmed influenza-illness caused by any antigenic subtype.

CONTACTS AND LOCATIONS:
Overall Officials: Pjt de Villiers, Professor, Principal Investigator — Dept of Family Medicine & Primary Care, University of Stellenbosch
Locations (1):
- Department of Family & Primary Care, Faculty of Medicine, University of Stellenbosch, Tygerberg, South Africa

REFERENCES:
- [Derived] De Villiers PJ, Steele AD, Hiemstra LA, Rappaport R, Dunning AJ, Gruber WC, Forrest BD; LAIV Elderly Study Trial Network. Efficacy and safety of a live attenuated influenza vaccine in adults 60 years of age and older. Vaccine. 2009 Dec 10;28(1):228-34. doi: 10.1016/j.vaccine.2009.09.092. Epub 2009 Sep 29. PMID 19796721